CLINICAL TRIAL: NCT03860935
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of AG10 in Subjects With Symptomatic Transthyretin Amyloid Cardiomyopathy (ATTRibute-CM Trial)
Brief Title: Efficacy and Safety of AG10 in Subjects With Transthyretin Amyloid Cardiomyopathy
Acronym: ATTRibute-CM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eidos Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG10-301; 2018-004280-32 (EudraCT Number)
Record Dates: First submitted 2019-02-27; First posted 2019-03-04 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Amyloidosis; Amyloid Cardiomyopathy; Transthyretin Amyloidosis; Cardiomyopathies; Heart Diseases
Keywords: Amyloidosis; ATTR-CM; Transthyretin; Amyloid; TTR
MeSH Terms: conditions — Amyloidosis; Amyloid Neuropathies, Familial; Amyloidosis, Hereditary, Transthyretin-Related; Cardiomyopathies; Heart Diseases; Alzheimer Disease | interventions — attruby

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- acoramidis HCl 800 mg (Experimental): Subjects will receive acoramidis HCl 800 mg twice daily. 6MWT primary outcome will be assessed at the end of 12 months. The hierarchical combination of All-Cause mortality, cumulative frequency of cardiovascular-related hospitalizations, change from baseline in NT-proBNP levels, and change from baseline in distance walked on the 6MWT will be assessed after 30 months of treatment.
  Interventions: Drug: acoramidis
- Placebo (Placebo Comparator): Subjects will receive placebo to match twice daily. 6MWT primary outcome will be assessed at the end of 12 months. The hierarchical combination of All-Cause mortality, cumulative frequency of cardiovascular-related hospitalizations, change from baseline in NT-proBNP levels, and change from baseline in distance walked on the 6MWT will be assessed after 30 months of treatment.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: acoramidis — TTR stabilizer administered orally twice daily (BID)
  Other Names: AG10; ALXN2060
  Arms: acoramidis HCl 800 mg
Drug: Placebo Oral Tablet — Non-active control administered orally twice daily (BID)
  Arms: Placebo

SUMMARY:
Phase 3 efficacy and safety study to evaluate acoramidis (AG10) HCl 800 mg administered orally twice a day compared to placebo in subjects with symptomatic Transthyretin Amyloid Cardiomyopathy (ATTR-CM).

DETAILED DESCRIPTION:
Transthyretin amyloid cardiomyopathy (ATTR-CM) is an underdiagnosed condition believed to affect more than 400,000 people worldwide. In ATTR-CM, the accumulation of transthyretin (TTR) amyloid results in thickening and stiffening of the heart, which often leads to heart failure or even death.

There are two forms of ATTR-CM:

* Wild Type* This form of the condition primarily develops in older individuals who do not carry gene mutations.
* Hereditary* This form of the condition comes from gene mutations passed down in families.

In this study we are researching the investigational drug acoramidis HCl 800 mg administered orally twice a day. Through the study, we want to evaluate the efficacy and safety of acoramidis in patients with ATTR-CM versus placebo.

This is a 30 month, randomized, double-blind, placebo-controlled study. This means that, during the 30 month study, investigators conducting the research and study participants will not know whether the study participant is receiving acoramidis or placebo.

The primary outcomes of the study are:

1. The impact of acoramidis versus placebo on the change in distance walked on the 6 minute walk test (6MWT) after 12 months of treatment compared to baseline.
2. The impact of acoramidis versus placebo on the hierarchical combination of All-Cause mortality, cumulative frequency of cardiovascular-related hospitalizations, change from baseline in NT-proBNP, and change in from baseline in 6MWT over a 30-month fixed treatment duration.

At the end of 30 months, participants may be eligible to receive investigational acoramidis, and there is no placebo. This is called an "open label extension." This separate study may help us better understand the safety related to taking acoramidis over a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

* Have an established diagnosis of ATTR-CM with either wild-type TTR or variant TTR genotype
* Have a history of heart failure evidenced by at least one prior hospitalization for heart failure or clinical evidence of heart failure without prior heart failure hospitalization manifested by signs or symptoms of volume overload or elevated intracardiac pressures or heart failure symptoms that required or require ongoing treatment with a diuretic.
* New York Heart Association (NYHA) Class I-III symptoms due to ATTR cardiomyopathy.
* On stable doses of cardiovascular medical therapy
* Completed ≥150 m on the 6MWT on 2 tests that are within 15% of total distance walked prior to randomization
* Biomarkers of myocardial wall stress, NT-proBNP level ≥300 pg/mL at screening
* Have left ventricular wall (interventricular septum or left ventricular posterior wall) thickness ≥12 mm

Exclusion Criteria:

* Had acute myocardial infarction, acute coronary syndrome or coronary revascularization, or experienced stroke or transient ischemic attack within 90 days prior to screening
* Has hemodynamic instability
* Likely to undergo heart transplantation within a year of screening
* Confirmed diagnosis of primary (light chain) amyloidosis
* Biomarkers of myocardial wall stress, NT-proBNP level ≥8500 pg/mL at screening
* Measure of kidney function, eGFR by MDRD formula <15 mL/min/1.73 m2
* Current treatment with marketed drug products and other investigational agents for the treatment of ATTR-CM
* Current treatment with calcium channel blockers with conduction system effects (e.g. verapamil, diltiazem). The use of dihydropyridine calcium channel blockers is allowed. The use of digitalis will only be allowed if required for management of atrial fibrillation with rapid ventricular response

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (103):
- United States (40):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Pacific Heart Institute, Santa Monica, California
  - University of Colorado Hospital - Anschutz Medical Campus, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Piedmont Heart Institute Athens, Athens, Georgia
  - Emory Heart and Vascular Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - MedStar Medical Group Cardiology at Franklin Square Medical Center, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Saint Elizabeth's Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - New York University Langone Health, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Laurelton Heart Specialist, Rosedale, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - The Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health - Greenville Memorial Hospital, Greenville, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Carilion Clinic Roanoke Heart Institute, Roanoke, Virginia
  - University of Washington School of Medicine, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
- Australia (6):
  - Royal Adelaide Hospital, Adelaide
  - Box Hill Hospital, Box Hill
  - Royal Hobart Hospital, Hobart
  - Fiona Stanley Hospital, Murdoch
  - Saint Vincent's Hospital Sydney, Sydney
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (5):
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk, Limburg
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt, Limburg
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende, Bruges, West Vlaanderen
  - Onze-Lieve-Vrouw Ziekenhuis Aalst, Aalst
  - Universitair Ziekenhuis Leuven, Leuven
- Brazil (5):
  - Hospital Cárdio Pulmonar, Salvador, Estado de Bahia
  - Santa Casa de Misericordia - Porto Alegre, Porto Alegre, Rio Grande do Sul
  - CAPED - Centro Avançado de Pesquisa e Estudos para o Diagnóstico, Ribeirão Preto, São Paulo
  - INCOR, São Paulo, São Paulo
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba - St. Boniface, Winnipeg, Manitoba
  - Halifax Infirmary, Halifax, Nova Scotia
  - Toronto Heart Centre, Toronto, Ontario
  - University of Toronto, Toronto, Ontario
  - Centre Hospitalier de L'Universite de Montreal - Hôpital Notre-Dame, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
  - Hôpital régional de Rimouski, Rimouski, Quebec
  - Montreal Heart Institute, Montreal
- Czechia (3):
  - St. Anne´s University Hospital, Brno-střed
  - General University Hospital in Prague, New Town
  - Institute for Clinical and Experimental Medicine, Prague
- Aarhus Universitetshospital, Aarhus, Dinamarca, Denmark
- Alexandra General Hospital of Athens, Athens, Attica, Greece
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - Saint Vincents University Hospital, Dublin
- Israel (2):
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (7):
  - Ospedale San Donato, Arezzo
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Toscana Gabriele Monasterio per la Ricerca Medica e di Sanità Pubblica, Pisa
  - Ospedale degli Infermi, Rimini
  - Universita degli Studi di Roma La Sapienza - Umberto I Policlinico di Roma, Roma
- Netherlands (3):
  - Maastricht Universitair Medisch Centrum, Maastricht, Limburg
  - Universitair Medisch Centrum Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht
- New Zealand (2):
  - Middlemore Hospital, Otahuhu, Auckland
  - Waikato Hospital, Hamilton, Waikato Region
- National Institute of Cardiology, Warsaw, Poland
- Portugal (2):
  - Centro Hospitalar de Lisboa Norte EPE- Hospital Santa Maria, Lisbon
  - Centro Hospitalar do Porto, Porto
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Gyeonggi-do
- Spain (8):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Juan Ramón Jiménez, Huelva
  - Clinica Universidad de Navarra Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Son Llàtzer, Palma de Mallorca
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (2):
  - Royal Free Hospital, London, England
  - Richmond Pharmacology, London

REFERENCES:
- [Derived] Gillmore JD, Judge DP, Cappelli F, Fontana M, Garcia-Pavia P, Gibbs S, Grogan M, Hanna M, Hoffman J, Masri A, Maurer MS, Nativi-Nicolau J, Obici L, Poulsen SH, Rockhold F, Shah KB, Soman P, Garg J, Chiswell K, Xu H, Cao X, Lystig T, Sinha U, Fox JC; ATTRibute-CM Investigators. A plain language review of the ATTRibute-CM study: efficacy and safety of acoramidis in transthyretin amyloid cardiomyopathy. Future Cardiol. 2025 Dec;21(12):1017-1025. doi: 10.1080/14796678.2025.2591426. Epub 2025 Dec 12. PMID 41384357
- [Derived] Alexander KM, Davis MK, Akinboboye O, Berk J, Bhatt K, Cappelli F, Cuddy SAM, Fontana M, Garcia-Pavia P, Gillmore JD, Griffin JM, Grodin JL, Judge DP, Khouri MG, Lam K, Masri A, Maurer MS, Obici L, Ruberg FL, Sarswat N, Shah K, Soman P, Stern L, Wright R, Xiong K, Cao X, Lystig T, Tamby JF, Castano A, Katz L, Sinha U, Fox JC, Solomon SD, Grogan M. Efficacy of Acoramidis in Wild-Type and Variant Transthyretin Amyloid Cardiomyopathy: Results From ATTRibute-CM and Its Open-Label Extension. JAMA Cardiol. 2026 Jan 1;11(1):57-67. doi: 10.1001/jamacardio.2025.4477. PMID 41205147
- [Derived] Dasgupta N, Poulsen SH, Emdin M, Ambardekar AV, Shah KB, Hennum L, Marwah R, Allison M, Shivanna P, Siddhanti S, Tamby JF, Falvey H, Grodin JL. Contemporary Oral Medication Use and Frequency in Patients with Transthyretin Amyloid Cardiomyopathy. Am J Cardiovasc Drugs. 2025 Nov;25(6):829-839. doi: 10.1007/s40256-025-00752-x. Epub 2025 Aug 1. PMID 40750720
- [Derived] Maurer MS, Judge DP, Gillmore JD, Garcia-Pavia P, Masri A, Cappelli F, Alexander KM, Sarswat N, Grogan M, Ambardekar AV, Ducharme A, Poulsen SH, Lam K, Obici L, Soman P, Rao S, Tamby JF, Castano A, Fox JC, Adam B, Chepyala SR, Poland B, Sinha U, Fontana M. Early Increase in Serum Transthyretin by Acoramidis Independently Predicts Improved Survival in TTR Amyloid Cardiomyopathy. J Am Coll Cardiol. 2025 May 27;85(20):1911-1923. doi: 10.1016/j.jacc.2025.03.542. PMID 40398971
- [Derived] Judge DP, Alexander KM, Cappelli F, Fontana M, Garcia-Pavia P, Gibbs SDJ, Grogan M, Hanna M, Masri A, Maurer MS, Obici L, Soman P, Cao X, Lystig T, Tamby JF, Siddhanti S, Castano A, Katz L, Fox JC, Mahaffey KW, Gillmore JD. Efficacy of Acoramidis on All-Cause Mortality and Cardiovascular Hospitalization in Transthyretin Amyloid Cardiomyopathy. J Am Coll Cardiol. 2025 Mar 18;85(10):1003-1014. doi: 10.1016/j.jacc.2024.11.042. PMID 40074465
- [Derived] Soman P, Khouri MG, Lenihan D, Reyentovich A, Sperry BW, Sowalsky K, Bai Y, Du J, Katz L, Siddhanti S, Fox JC. Comparison of in-clinic assessment of 6MWT by conventional method and using wearable sensors for patients with ATTR-CM. Future Cardiol. 2025 Feb;21(2):75-81. doi: 10.1080/14796678.2025.2457881. Epub 2025 Jan 29. PMID 39878480
- [Derived] Gillmore JD, Judge DP, Cappelli F, Fontana M, Garcia-Pavia P, Gibbs S, Grogan M, Hanna M, Hoffman J, Masri A, Maurer MS, Nativi-Nicolau J, Obici L, Poulsen SH, Rockhold F, Shah KB, Soman P, Garg J, Chiswell K, Xu H, Cao X, Lystig T, Sinha U, Fox JC; ATTRibute-CM Investigators. Efficacy and Safety of Acoramidis in Transthyretin Amyloid Cardiomyopathy. N Engl J Med. 2024 Jan 11;390(2):132-142. doi: 10.1056/NEJMoa2305434. PMID 38197816
- [Derived] Stern LK, Kittleson MM. Updates in Cardiac Amyloidosis Diagnosis and Treatment. Curr Oncol Rep. 2021 Mar 16;23(4):47. doi: 10.1007/s11912-021-01028-8. PMID 33725199

RESULTS

PARTICIPANT FLOW:
Groups:
- Acoramidis HCl 800 mg: Participants with symptomatic ATTR-CM received 800 mg acoramidis HCl BID (two 400 mg acoramidis HCl tablets, each equivalent to 356 mg acoramidis [active moiety])
- Placebo: Participants with symptomatic ATTR-CM received matching placebo (two matching placebo tablets BID)
Period: Overall Study
Arm/Group | Acoramidis HCl 800 mg | Placebo
Started | 421 | 211
Completed | 331 | 154
Not Completed | 90 | 57
Not completed — Withdrawal of Consent | 15 | 6
Not completed — Death | 75 | 51

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Acoramidis HCl 800 mg | Placebo | Total
Number analyzed (Participants) | 421 | 211 | 632
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 9 | 21
  >=65 years | 409 | 202 | 611
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.37 (6.450) | 77.09 (6.763) | 77.27 (6.552)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 25 | 62
  Male | 384 | 186 | 570
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 401 | 199 | 600
  Unknown or Not Reported | 12 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 10 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 20 | 10 | 30
  White | 368 | 187 | 555
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 21 | 9 | 30
Distance Walked During the 6 Minute Walk Test (6MWT) [Mean (Standard Deviation); unit: Meter] — Secondary Outcome Measure at Baseline Population: Participants evaluable by each baseline assessment.
  Meter
    number analyzed (Participants) | 419 | 211 | 630
    (all) | 361.21 (103.705) | 348.37 (93.564) | 356.91 (100.531)
Kansas City Cardiomyopathy Questionnaire Overall Score (KCCQ-OS) [Mean (Standard Deviation); unit: units on a scale] — Secondary Outcome Measure at Baseline Population: Participants evaluable by each baseline assessment
  units on a scale
    number analyzed (Participants) | 420 | 211 | 631
    (all) | 71.52 (19.387) | 70.31 (20.541) | 71.12 (19.773)
Serum TTR (Prealbumin) Level [Mean (Standard Deviation); unit: mg/dL] — Secondary Outcome Measure at Baseline Population: Participants evaluable by each baseline assessment
  mg/dL
    number analyzed (Participants) | 418 | 208 | 626
    (all) | 23.16 (5.643) | 23.63 (6.070) | 23.32 (5.788)

OUTCOME MEASURES:

1. Primary Outcome: A Hierarchical Combination of All-Cause Mortality, Cumulative Frequency of CV-related Hospitalization, Change From Baseline in NT-proBNP and Change From Baseline in 6MWT at the Last Available Visit Where Both Subjects Had Non-missing Assessments.
Description: The endpoint was analyzed using Finkelstein-Schoenfeld method. The method combines all-cause mortality, cumulative frequency of CV-related hospitalizations, change from baseline in NT-proBNP and change from baseline in 6MWT in a hierarchical fashion. The method compares every participant with every other participant within strata, assigning a +1 to the "better" participant and a -1 to the "worse" participant and 0 if they are "tied". Participants who had heart transplantation or implantation of a cardiac mechanical assist device were handled in the same manner as death. 'Win' represents a participant doing better based on hierarchical comparison. The reported unit is the total percent of "wins" for each treatment group from performing such a hierarchical comparison across stratification factors in the study.
Time Frame: Baseline up to Month 30
Population: The mITT population includes subjects who meet the definition of ITT which includes all randomized subjects who received at least one dose of IMP and have at least one post baseline efficacy assessment as well as an additional requirement which is to have a baseline eGFR >= 30 mL/min/1.73 m^2 . Subjects in this population were analyzed according to their assigned randomized treatment.
Measure: Number; unit: Percent of Wins from Win Ratio
Arm/Group | Acoramidis HCl 800 mg | Placebo
Number analyzed (Participants) | 409 | 202
Percent of Wins from Win Ratio | 63.7 | 35.9
Statistical Analysis 1: Comparison: Acoramidis HCl 800 mg vs Placebo; Test type: Superiority; p < 0.0001, Finkelstein-Schoenfeld Method

2. Secondary Outcome: Change From Baseline to Month 30 in the Distance Walked During the 6 Minute Walk Test (6MWT)
Description: 6MWT measures the total distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed.
Time Frame: Month 30
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Meter
Arm/Group | Acoramidis HCl 800 mg | Placebo
Number analyzed (Participants) | 384 | 186
Meter | -64.65 (5.508) | -104.29 (7.772)
Statistical Analysis 1: Comparison: Acoramidis HCl 800 mg vs Placebo; LS means are from a MMRM model with treatment group, visit, randomization stratification factors of genotype, NT-proBNP level and eGFR level (as recorded in IXRS) and treatment group-by-visit interaction as factors, and baseline value as covariate. Missing measurements due to early discontinuation of study treatment and due to death were imputed using the Jump to Reference (J2R) method and sampling with replacement from the worst 5% of observed values, respectively, as specified in study SAP; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = 39.64, 96% CI 2-sided [20.18 to 59.10], Standard Error of Mean 9.477

3. Secondary Outcome: Change From Baseline to Month 30 of the Kansas City Cardiomyopathy Questionnaire Overall Score (KCCQ-OS)
Description: KCCQ is a 23-item participant-completed questionnaire that assesses health status and health-related quality of life in participants with heart failure. Eight domain scores were calculated for the KCCQ: Physical limitation, Social limitation, Quality of life, Self-efficacy, Symptom stability, Symptom frequency, Symptom burden, and Total symptoms (calculated as the mean of Symptom frequency and Symptom burden scores). The summary score of Overall Summary (calculated as mean of Physical limitation, Social limitation, Total symptoms, and Quality of life scores) was calculated. Domain and summary scores were scaled to range from 0 (minimum) to 100 (maximum); higher scores represent better health status.
Time Frame: Month 30
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Acoramidis HCl 800 mg | Placebo
Number analyzed (Participants) | 405 | 201
Score on a scale | -11.48 (1.181) | -21.42 (1.651)
Statistical Analysis 1: Comparison: Acoramidis HCl 800 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = 9.94, 96% CI 2-sided [5.79 to 14.10], Standard Error of Mean 2.024

4. Secondary Outcome: Change From Baseline to Month 30 in Serum TTR (Prealbumin) Level
Description: Serum TTR (Prealbumin) is an in vivo biomarker of stabilization.
Time Frame: Month 30
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Acoramidis HCl 800 mg | Placebo
Number analyzed (Participants) | 397 | 197
mg/dL | 5.78 (0.391) | -1.32 (0.541)
Statistical Analysis 1: Comparison: Acoramidis HCl 800 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares Mean Difference = 7.10, 96% CI 2-sided [5.73 to 8.46], Standard Error of Mean 0.665

5. Secondary Outcome: All-cause Mortality by Month 30, Including Death Due to Any Cause, Heart Transplant or Cardiac Mechanical Assist Device (CMAD)
Description: Number of deaths due to any cause was analyzed. Participants who had heart transplantation or implantation of a CMAD were handled in the same manner as death.
Time Frame: Baseline up to Month 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Acoramidis HCl 800 mg | Placebo
Number analyzed (Participants) | 409 | 202
Participants | 79 | 52
Statistical Analysis 1: Comparison: Acoramidis HCl 800 mg vs Placebo; Test type: Superiority; p = 0.0569, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test is stratified by randomization stratification factors of genotype, NT-proBNP level and eGFR level as recorded in IXRS; Relative Risk Reduction (%) = 25

ADVERSE EVENTS:
Time Frame: In Study AG10-301 participants, treatment emergent adverse events (TEAEs) are defined as (a) events with onset after the first dose of study drug, or (b) if the event was present before the first dose of study drug, but increased in severity after the first dose of study drug, and (c) with onset date or severity increase date <= 30 days after the last dose of study drug (through AG10-301 Study completion, 30 months) or until the first dose in open label extension Study AG10-304.
Description: Study AG10-301 TEAEs are any untoward or unfavorable medical occurrence in a participant, whether or not considered related to the participant's participation in the research, with event onset date or increase in severity date as defined in the Time Frame Section above. Serious TEAEs and non-serious TEAEs are also presented separately below.
Arm/Group | Acoramidis HCl 800 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 84/421 | 55/211
Serious Adverse Events (participants affected / at risk) | 230/421 | 137/211
Other Adverse Events (participants affected / at risk) | 410/421 | 199/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acoramidis HCl 800 mg (N=421) | Placebo (N=211)
Cardiac failure (Cardiac disorders) | 45 | 39
Cardiac failure acute (Cardiac disorders) | 21 | 14
Atrial fibrillation (Cardiac disorders) | 19 | 15
Bradycardia (Cardiac disorders) | 11 | 2
Ventricular tachycardia (Cardiac disorders) | 6 | 5
Atrioventricular block complete (Cardiac disorders) | 8 | 3
Acute myocardial infarction (Cardiac disorders) | 5 | 4
Cardiac failure chronic (Cardiac disorders) | 6 | 3
Cardiac arrest (Cardiac disorders) | 4 | 4
Cardiac failure congestive (Cardiac disorders) | 5 | 3
Cardiorenal syndrome (Cardiac disorders) | 3 | 3
Atrial flutter (Cardiac disorders) | 3 | 3
Acute left ventricular failure (Cardiac disorders) | 3 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 3
Atrioventricular block (Cardiac disorders) | 2 | 2
Cardiac amyloidosis (Cardiac disorders) | 2 | 2
Angina pectoris (Cardiac disorders) | 2 | 1
Right ventricular failure (Cardiac disorders) | 1 | 2
Sinus node dysfunction (Cardiac disorders) | 3 | 0
Trifascicular block (Cardiac disorders) | 2 | 1
Atrial tachycardia (Cardiac disorders) | 2 | 0
Chronic left ventricular failure (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Bifascicular block (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bundle branch block (Cardiac disorders) | 1 | 0
Cardiac flutter (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 12 | 6
COVID-19 (Infections and infestations) | 9 | 4
Urinary tract infection (Infections and infestations) | 7 | 3
COVID-19 pneumonia (Infections and infestations) | 2 | 8
Cellulitis (Infections and infestations) | 7 | 3
Sepsis (Infections and infestations) | 4 | 2
Septic shock (Infections and infestations) | 4 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Erysipelas (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 2 | 1
Abscess limb (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Pneumonia aspiration (Infections and infestations) | 2 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1
Post procedural infection (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0
Infective tenosynovitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Sepsis pasteurella (Infections and infestations) | 0 | 1
Septic arthritis streptococcal (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin graft infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 13 | 2
Rib fracture (Injury, poisoning and procedural complications) | 5 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Eschar (Injury, poisoning and procedural complications) | 1 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 6 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 3 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal metaplasia (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 6 | 4
Presyncope (Nervous system disorders) | 5 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 2
Cerebral infarction (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 1 | 1
Embolic stroke (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Chorea (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Cranial nerve paralysis (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 21 | 8
Haematuria (Renal and urinary disorders) | 3 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 2
Renal impairment (Renal and urinary disorders) | 3 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
End stage renal disease (Renal and urinary disorders) | 1 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Death (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 2 | 2
Chest pain (General disorders) | 1 | 2
Asthenia (General disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 0
Complication associated with device (General disorders) | 1 | 0
Cyst (General disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 3 | 4
Aortic stenosis (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 3 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Femoral artery embolism (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Varicose vein ruptured (Vascular disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 7 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Cardiac output decreased (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1
Troponin T increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura senile (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Device failure (Product Issues) | 1 | 0
Device loosening (Product Issues) | 1 | 0
Device malfunction (Product Issues) | 0 | 1
Lead dislodgement (Product Issues) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Macular hole (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Amyloidosis (Immune system disorders) | 0 | 1
Euthanasia (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acoramidis HCl 800 mg (N=421) | Placebo (N=211)
COVID-19 (Infections and infestations) | 80 | 27
Urinary tract infection (Infections and infestations) | 46 | 26
Upper respiratory tract infection (Infections and infestations) | 22 | 12
Nasopharyngitis (Infections and infestations) | 21 | 11
Constipation (Gastrointestinal disorders) | 51 | 31
Diarrhoea (Gastrointestinal disorders) | 48 | 16
Nausea (Gastrointestinal disorders) | 24 | 11
Abdominal pain upper (Gastrointestinal disorders) | 22 | 3
Cardiac failure (Cardiac disorders) | 69 | 61
Atrial fibrillation (Cardiac disorders) | 55 | 36
Ventricular tachycardia (Cardiac disorders) | 12 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 34 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 11
Dizziness (Nervous system disorders) | 45 | 22
Syncope (Nervous system disorders) | 15 | 12
Gout (Metabolism and nutrition disorders) | 46 | 17
Hypervolaemia (Metabolism and nutrition disorders) | 21 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 11
Decreased appetite (Metabolism and nutrition disorders) | 19 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 7
Fatigue (General disorders) | 42 | 26
Oedema peripheral (General disorders) | 33 | 25
Asthenia (General disorders) | 21 | 8
Peripheral swelling (General disorders) | 6 | 14
Fall (Injury, poisoning and procedural complications) | 59 | 38
Skin laceration (Injury, poisoning and procedural complications) | 11 | 11
Blood creatinine increased (Investigations) | 26 | 4
Weight decreased (Investigations) | 16 | 13
Renal impairment (Renal and urinary disorders) | 35 | 17
Acute kidney injury (Renal and urinary disorders) | 35 | 16
Haematuria (Renal and urinary disorders) | 17 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 8
Rash (Skin and subcutaneous tissue disorders) | 21 | 11
Hypotension (Vascular disorders) | 30 | 14
Insomnia (Psychiatric disorders) | 20 | 15
Anaemia (Blood and lymphatic system disorders) | 33 | 15
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT03860935/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT03860935/SAP_001.pdf